CLINICAL TRIAL: NCT06363487
Title: Effects of Single-dose Semaglutide on Cognition and Energy in Healthy Volunteers
Brief Title: Semaglutide and Cognition in Healthy Volunteers
Acronym: OxSENSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: R87970/RE001
Record Dates: First submitted 2024-04-09; First posted 2024-04-12 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2024-04

CONDITIONS: Cognitive Change
Keywords: Semaglutide; Healthy volunteers; Experimental medicine; Cognition; Reward; Emotional processing; Memory; Energy
MeSH Terms: interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Semaglutide (Experimental): Semaglutide pre-filled pen, 0.5mg in 1.5mL, subcutaneous injection
  Interventions: Drug: Semaglutide, 0.5 mg/mL
- Placebo (Placebo Comparator): Saline solution 0.9% NaCl, solution for injection 1.5mL, subcutaneous injection syringe
  Interventions: Other: Placebo, 0.9% NaCl 1.5mL

INTERVENTIONS:
Drug: Semaglutide, 0.5 mg/mL — Injected subcutaneously (pre-filled pen) in the upper arm (preferred site), in the abdomen, or in the thigh according to participant's preference. The participant will be asked to wear an eye blindfold during the time of the study medication/placebo administration, to avoid compromising blinding. It is not possible to blind the researcher administering the medication/placebo because semaglutide comes in specific pre-filled pens. The person who administers the subcutaneous injection will be suitably trained and experienced, and have been authorised to do so by the Principal Investigator - they will not be involved in other aspects of the study for that participant to avoid compromising blinding.
  Arms: Semaglutide
Other: Placebo, 0.9% NaCl 1.5mL — Injected subcutaneously (subcutaneous injection syringe) in the upper arm (preferred site), in the abdomen, or in the thigh according to participant's preference. The participant will be asked to wear an eye blindfold during the time of the study medication/placebo administration, to avoid compromising blinding. The person who administers the subcutaneous injection will be suitably trained and experienced, and have been authorised to do so by the Principal Investigator - they will not be involved in other aspects of the study for that participant to avoid compromising blinding.
  Arms: Placebo

SUMMARY:
Semaglutide is a glucagon-like peptide 1 receptor agonist (GLP-1RA). It is a safe medication approved for use in type-2 diabetes mellitus (T2DM) and obesity. Primarily, it works by counteracting insulin-resistance and inducing weight loss. It also acts on several other interconnected neurobiological, immunological (esp. inflammatory), endocrine-metabolic, and gut-brain axis processes that play a role in depressive symptoms. Its effects on cognition and energy are currently unknown. In this study we are using semaglutide as an experimental tool to further investigate these relationships.

DETAILED DESCRIPTION:
Semaglutide is a novel GLP-1RA licensed for T2DM and obesity, which mainly works by offsetting insulin-resistance and stimulating weight loss (1). It also acts on various neurobiological, immunological, endocrine-metabolic, and gut-brain axis processes that play a role in depressive symptoms (2). Preliminary evidence suggests these drugs are safe from a neuropsychiatric perspective (3) and could be beneficial in unipolar (4) and bipolar depression (5) - an outcome possibly mediated by inflammatory pathways (6).

The proposed study investigates the effects of semaglutide on cognition and energy, which are currently unknown. Work in our laboratory established that short-term use of conventional antidepressants in healthy volunteers shifts reward sensitivity and emotional cognition (7) - an important neuropsychological mechanism of antidepressant action (8). An experimental medicine trial that assesses the effects of semaglutide on reward sensitivity emotional cognition can validate its potential to be repurposed for treating depressive disorders (9). Moreover, brain insulin resistance, likely lessened by semaglutide, is associated with deficit in impulse-control as well as non-emotional cognitive and energy impairment in people with depression (10). Finally, defining the overall cognitive and energy profile of semaglutide is important for the many people already taking it for its licensed indications (i.e., T2DM, obesity).

Therefore, the primary objective of this study is to assess the effect of a single dose of semaglutide 0.5mg subcutaneous injection vs placebo on reward sensitivity tasks in healthy volunteers. Secondary objectives include the investigation of the effects of semaglutide on other cognitive domains (emotional processing, impulsivity, memory) and energy/activity levels. Psychological questionnaires are also measured as relevant covariates.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Aged from 21 to 55 years
* Body Mass Index (BMI) from 18 to 30 (because our main outcomes involve cognitive and energy measures, this decision regarding the BMI range has been taken with the purpose of including a more homogeneous sample of healthy participants in terms of baseline cognitive and energy levels)
* Sufficiently fluent English to understand and complete the tasks
* Participant is willing and able to give informed consent for participation in the research
* Not currently taking any regular medications (except the contraceptive pill)

Exclusion Criteria:

* Currently on any regular prescribed medications (except the contraceptive pill), unless unlikely to compromise safety or affect data quality in the opinion of the medical supervisor according to clinical judgement
* History of, or current significant psychiatric illness in the opinion of the medical supervisor according to clinical judgement
* Current alcohol or substance misuse disorder (<6 months)
* Current moderate or severe dyslexia
* History of, or current significant medical illness in the opinion of the medical supervisor according to clinical judgement
* History of, or current pancreatitis
* History of, or current severe congestive heart failure, end-stage renal disease, hepatic disease
* History of, or current significant neurological condition (e.g., epilepsy)
* History of, or current significant thyroid disorder
* History (including family history) of, or current multiple endocrine neoplasia syndrome type-2 (MEN 2) or medullary thyroid carcinoma (MTC)
* Known type-1 or type-2 diabetes mellitus
* Known hypersensitivity to the study drug (i.e., semaglutide)
* Pregnant, breast feeding, or person of child-bearing potential not using appropriate contraceptive measures including hormonal contraception, intrauterine device, bilateral tubal occlusion, vasectomised partner, condom, absolute sexual abstinence - periodic sexual abstinence, withdrawal, and spermicides-only are not acceptable methods of contraception
* Participation in a study that uses the same or similar computer tasks (O-ETB, see below) as those used in the present study
* Participation in a study that involves the use of a medication within the last 3 months

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2024-06-06 (Actual); Primary Completion 2024-12-11 (Actual); Study Completion 2024-12-11 (Actual)

PRIMARY OUTCOMES:
Reward (learning) | 6-7 days
  Win/loss and valence on a computer-based task of reward processing (i.e., probabilistic instrumental learning task), comparing those receiving drug vs placebo.
Reward (effort-based) | 6-7 days
  Win/loss and valence on a computer-based task of reward processing (i.e., apple-gathering task), comparing those receiving drug vs placebo.
Reward (primary) | 6-7 days
  Valence on a computer-based task of reward processing (i.e., taste strip task), comparing those receiving drug vs placebo.

SECONDARY OUTCOMES:
Emotional processing | 6-7 days
  Accuracy and reaction times on a computer-based task of emotional processing (i.e., facial expression recognition), comparing those receiving drug vs placebo.
Emotional impulsivity | 6-7 days
  Accuracy and reaction times on a computer-based task of emotional response inhibition (i.e., affective go/no-go task), comparing those receiving drug vs placebo.
Memory (short- and medium-term) processing | 6-7 days
  Accuracy and reaction times on a computer-based tasks of (short- and medium-term) memory (auditory-verbal learning task), comparing those receiving drug vs placebo.
Memory (working) processing | 6-7 days
  Accuracy and reaction times on a computer-based task of working memory (N-back), comparing those receiving drug vs placebo.
Energy/activity | Across 6-7 days
  Ecological momentary assessment (4 times/day) on 7-point Likert energy/activity scale (very tired to very energetic, very inactive to very active)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry, University of Oxford, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Anonymised research data without any personal data (e.g., reaction time data) will also be stored on private Open Science Framework (OSF) project components that are accessible only to the research team. We have previously confirmed with the University's Sponsor (formerly CTRG) in December 2019 that OSF can be used in this way to store anonymised data (with no personal data or linking files). Parts of the data might be uploaded to online data repositories or made publicly available on OSF in a completely anonymised fashion, to facilitate open science. Data uploaded in this way will be stored on OSF indefinitely.

REFERENCES:
- [Background] Collins L, Costello RA. Glucagon-Like Peptide-1 Receptor Agonists. 2024 Feb 29. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK551568/ PMID 31855395
- [Background] Detka J, Glombik K. Insights into a possible role of glucagon-like peptide-1 receptor agonists in the treatment of depression. Pharmacol Rep. 2021 Aug;73(4):1020-1032. doi: 10.1007/s43440-021-00274-8. Epub 2021 May 18. PMID 34003475
- [Background] O'Neil PM, Aroda VR, Astrup A, Kushner R, Lau DCW, Wadden TA, Brett J, Cancino AP, Wilding JPH; Satiety and Clinical Adiposity - Liraglutide Evidence in individuals with and without diabetes (SCALE) study groups. Neuropsychiatric safety with liraglutide 3.0 mg for weight management: Results from randomized controlled phase 2 and 3a trials. Diabetes Obes Metab. 2017 Nov;19(11):1529-1536. doi: 10.1111/dom.12963. Epub 2017 Jul 21. PMID 28386912
- [Background] Pozzi M, Mazhar F, Peeters GGAM, Vantaggiato C, Nobile M, Clementi E, Radice S, Carnovale C. A systematic review of the antidepressant effects of glucagon-like peptide 1 (GLP-1) functional agonists: Further link between metabolism and psychopathology: Special Section on "Translational and Neuroscience Studies in Affective Disorders". Section Editor, Maria Nobile MD, PhD. This Section of JAD focuses on the relevance of translational and neuroscience studies in providing a better understanding of the neural basis of affective disorders. The main aim is to briefly summaries relevant research findings in clinical neuroscience with particular regards to specific innovative topics in mood and anxiety disorders. J Affect Disord. 2019 Oct 1;257:S0165-0327(19)30593-2. doi: 10.1016/j.jad.2019.05.044. Epub 2019 May 28. PMID 31153593
- [Background] Mansur RB, Ahmed J, Cha DS, Woldeyohannes HO, Subramaniapillai M, Lovshin J, Lee JG, Lee JH, Brietzke E, Reininghaus EZ, Sim K, Vinberg M, Rasgon N, Hajek T, McIntyre RS. Liraglutide promotes improvements in objective measures of cognitive dysfunction in individuals with mood disorders: A pilot, open-label study. J Affect Disord. 2017 Jan 1;207:114-120. doi: 10.1016/j.jad.2016.09.056. Epub 2016 Oct 1. PMID 27721184
- [Background] Moulton CD, Pickup JC, Amiel SA, Winkley K, Ismail K. Investigating incretin-based therapies as a novel treatment for depression in type 2 diabetes: Findings from the South London Diabetes (SOUL-D) Study. Prim Care Diabetes. 2016 Apr;10(2):156-9. doi: 10.1016/j.pcd.2015.06.003. Epub 2015 Jun 29. PMID 26137918
- [Background] Harmer CJ, Shelley NC, Cowen PJ, Goodwin GM. Increased positive versus negative affective perception and memory in healthy volunteers following selective serotonin and norepinephrine reuptake inhibition. Am J Psychiatry. 2004 Jul;161(7):1256-63. doi: 10.1176/appi.ajp.161.7.1256. PMID 15229059
- [Background] Harmer CJ, Duman RS, Cowen PJ. How do antidepressants work? New perspectives for refining future treatment approaches. Lancet Psychiatry. 2017 May;4(5):409-418. doi: 10.1016/S2215-0366(17)30015-9. Epub 2017 Jan 31. PMID 28153641
- [Background] Godlewska BR, Harmer CJ. Cognitive neuropsychological theory of antidepressant action: a modern-day approach to depression and its treatment. Psychopharmacology (Berl). 2021 May;238(5):1265-1278. doi: 10.1007/s00213-019-05448-0. Epub 2020 Jan 15. PMID 31938879
- [Background] Hamer JA, Testani D, Mansur RB, Lee Y, Subramaniapillai M, McIntyre RS. Brain insulin resistance: A treatment target for cognitive impairment and anhedonia in depression. Exp Neurol. 2019 May;315:1-8. doi: 10.1016/j.expneurol.2019.01.016. Epub 2019 Jan 26. PMID 30695707
- [Background] Pessiglione M, Seymour B, Flandin G, Dolan RJ, Frith CD. Dopamine-dependent prediction errors underpin reward-seeking behaviour in humans. Nature. 2006 Aug 31;442(7106):1042-5. doi: 10.1038/nature05051. Epub 2006 Aug 23. PMID 16929307
- [Background] Bonnelle V, Veromann KR, Burnett Heyes S, Lo Sterzo E, Manohar S, Husain M. Characterization of reward and effort mechanisms in apathy. J Physiol Paris. 2015 Feb-Jun;109(1-3):16-26. doi: 10.1016/j.jphysparis.2014.04.002. Epub 2014 Apr 18. PMID 24747776
- [Background] Amsterdam JD, Settle RG, Doty RL, Abelman E, Winokur A. Taste and smell perception in depression. Biol Psychiatry. 1987 Dec;22(12):1481-5. doi: 10.1016/0006-3223(87)90108-9. No abstract available. PMID 3676376
- [Background] Harmer CJ, O'Sullivan U, Favaron E, Massey-Chase R, Ayres R, Reinecke A, Goodwin GM, Cowen PJ. Effect of acute antidepressant administration on negative affective bias in depressed patients. Am J Psychiatry. 2009 Oct;166(10):1178-84. doi: 10.1176/appi.ajp.2009.09020149. Epub 2009 Sep 15. PMID 19755572
- [Background] Colwell, M. J., Murphy, S., & Harmer, C. J. (2022). Emotional Go/No-Go Task (Oxford) (Psychopy). Zenodo. https://doi.org/10.5281/zenodo.6207865
- [Background] KIRCHNER WK. Age differences in short-term retention of rapidly changing information. J Exp Psychol. 1958 Apr;55(4):352-8. doi: 10.1037/h0043688. No abstract available. PMID 13539317
- [Background] Halahakoon DC, Kaltenboeck A, Martens M, Geddes JG, Harmer CJ, Cowen P, Browning M. Pramipexole Enhances Reward Learning by Preserving Value Estimates. Biol Psychiatry. 2024 Feb 1;95(3):286-296. doi: 10.1016/j.biopsych.2023.05.023. Epub 2023 Jun 15. PMID 37330165